CLINICAL TRIAL: NCT02040688
Title: Sensory Integration (Processing) Disorder Among Children With Behavioral Insomnia and Children With Feeding Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-11-RT-0471-11-CTIL
Record Dates: First submitted 2014-01-09; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: SID; Feeding Disorder; SPD
MeSH Terms: conditions — Sudden Infant Death; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Sleep Disorders: 7-36 months old children with behavioral insomnia of childhood based on the International Classification of Sleep Disorders (ICSD) criteria will be recruited from the Pediatric Sleep Center at Dana Children's hospital
- Control: 7-36 months old chidren of age who attend well-care clinics in the metropolitan of Tel Aviv for routine periodic medical examination.
- Feeding disorder: 7-36 monthsold children with feeding disorders based on Chatoor criteria will be recruited from the clinic of feeding disorders at Dana Children's Hospital.

SUMMARY:
Behavioral insomnia of childhood is a prevalent condition, affecting 10-30% of children 6-36 months of age. If left untreated, bedtime problems and night wakings can negatively impact the daytime functioning and behavior of the child, as well as the entire family.

Feeding difficulties are common in pediatric practice and encompass a spectrum ranging from children with physiological difficulties in ingesting food, through picky eaters to full fledged infantile feeding disorders.

We have recently shown that feeding and eating difficulties are more prevalent among children with behavioral insomnia of childhood and that sleep problems are more frequent in children with feeding disorders.

We hypotesize that SPD is a common etiology for both sleep and feeding disorders and that children with sleep or feeding disorder have increased rate of Sensory intergration disorder (SID) compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* children 7-36 months of age with behavioral insomnia of childhood based on the International Classification of Sleep Disorders (ICSD) criteria .
* children 7-36 months of age with feeding disorders based on Chatoor criteria.
* children 7-36 months of age who attend well-care clinics in the metropolitan of Tel Aviv for routine periodic medical examination.

Exclusion Criteria:

Children with

* Chronic medical conditions.
* Congenital abnormalities.
* Significant developmental delay.

Ages: 7 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 7-36 months old children will be selected from:
  * The clinic of feeding disorders at Dana Children's Hospital.
  * The Pediatric Sleep Center at Dana Children's hospital
  * Well-care clinics in the metropolitan of Tel Aviv
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sleep disorders using Brief Infant Sleep Questionnaire (BISQ) and feeding disorders using the Behavioral Pediatrics Feeding Assessment. | Imidietly after the questionnaire filled by the parent.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Sleep Center at Dana Children's hospital, Tel Aviv, Israel